CLINICAL TRIAL: NCT03524170
Title: RACHEL1: A Phase I Radiation and Checkpoint Blockade Trial in Patients With Metastatic Hormone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: Radiation Therapy and M7824 in Treating Patients With Metastatic Hormone Receptor Positive, HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0499; NCI-2018-00961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0499 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — bintrafusp alfa protein, human; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (M7824, radiation therapy) (Experimental): Patients receive M7824 IV over 1 hour every 14 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Beginning within 3 days after second dose of M7824, patients undergo radiation therapy QD for 5-10 days depending on the site of disease in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of anti-PD-L1/TGFbetaRII fusion protein M7824 (M7824) when given together with radiation therapy in treating patients with hormone receptor positive, HER2 negative breast cancer that has spread to other parts of the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. M7824 is a drug that targets specific proteins on immune cells in order to activate immune responses against tumor cells. Giving M7824 together with radiation therapy may work better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of M7824 and radiation therapy in patients with metastatic hormone receptor positive (HR+)/HER2 negative (-) breast cancer.

II. To evaluate the safety and tolerability of M7824 and radiation therapy in patients with metastatic HR+/HER2- breast cancer.

SECONDARY OBJECTIVES:

I. To assess immunologic/molecular responses, specifically percentage (%) change in tumor-infiltrating lymphocytes (TIL) pre and post therapy to M7824 and radiation therapy in patients with HR+/HER2- metastatic breast cancer.

II. To explore progression free survival (PFS) and overall survival (OS) to power future definitive trial.

III. To evaluate the in-field and abscopal effect of treatment with anti-PD-L1/TGF-beta trap (M7824) and radiation therapy.

EXPLORATORY OBJECTIVES:

I. To characterize the effect of anti-PD-L1/TGF-beta trap (M7824) and radiation therapy on immune biomarkers including PD-L1 expression and fibrosis changes in tumor microenvironment in tumor tissue obtained from subjects pre- and post-treatment.

II. To characterize circulating immune cell populations and cytokine profiles in tumor and circulation following treatment with M7824.

III. To conduct ribonucleic acid sequencing (RNAseq), RNA Scope, whole exome sequencing (WES) targeted sequencing and tissue IO gene expression.

OUTLINE:

Patients receive M7824 intravenously (IV) over 1 hour every 14 days. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Beginning within 3 days after second dose of M7824, patients undergo radiation therapy once a day (QD) for 5-10 days depending on the site of disease in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial and has signed the appropriate written informed consent form, approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the performance of any trial activities.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Highly effective contraception for both male and female subjects if the risk of conception exists. Highly effective contraception must be used 30 days prior to first trial administration, for the duration of trial treatment, and at least for 4 months after stopping trial treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately.
* Has confirmed HR+ and HER2 negative breast cancer with known metastatic disease. HR defined as positive if expression greater than 10% by immunohistochemistry (IHC). HER2 negative or non-amplified is determined by the current American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) criteria which are as follows: HER2 testing by IHC as 0 or 1+. If HER2 is 2+, ISH (in situ hybridization) must be performed. HER2 is positive if: i. IHC 3+ based on circumferential membrane staining that is a. complete, intense ii. ISH positive based on: a. single-probe average HER2 copy number >= 6.0 signals/cell. b. Dual-probe HER2/CEP17 ratio >= 2.0 with an average HER2 copy number >= 4.0 signals/cell c. Dual-probe HER2/CEP17 ratio >= 2.0 with an average HER2 copy number < 4.0 signals/cell d. Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number >= 6.0 signals/cell.
* Has at least 2 identified sites of metastatic disease by imaging.
* Has received no more than 5 previous lines of chemotherapy and has received at least one line of therapy with an endocrine therapy or endocrine therapy combination.
* White blood cell (WBC) count >= 3 x 10^9/L.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L.
* Lymphocyte count >= 0.5 x 10^9/L.
* Platelet count >= 100 x 10^9/L.
* Hemoglobin (Hgb) >= 9 g/dL.
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN).
* Aspartate aminotransferase (AST) level =< 2.5 x ULN.
* Alanine aminotransferase (ALT) level =< 2.5 x ULN.
* International normalized ratio (INR) < 1.5.
* Adequate renal function defined by an estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula or be measure for creatinine clearance from 24 hour urine collection.
* Has not had major surgery within 28 days prior to starting study treatment. Central venous access surgeries and/or placements would not be considered as major surgery.
* Is eligible for palliative radiotherapy as determined by the treating radiation oncologist.

Exclusion Criteria:

* Anticancer treatment within 14 days before the start of trial treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative radiotherapy delivered in a normal organ-sparing technique], immune therapy, or cytokine therapy).
* Major surgery as determined by the investigator within 28 days before the start of trial treatment (prior diagnostic biopsy is permitted).
* Systemic therapy with immunosuppressive agents within 7 days before the start of treatment; or use of any investigational drug within 28 days before the start of trial treatment.
* Subjects with active central nervous system (CNS) metastases with significant neurological compromise or symptoms are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy), who show no evolving new neurological symptoms are eligible for the study.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
* Significant acute or chronic infections including, among others: a. Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. b. Active hepatitis B virus (HBV) (HBV surface antigen positive) or hepatitis C virus (HCV) (HCV RNA positive). c. Subjects with known active tuberculosis (history of exposure or history of positive tuberculosis test plus presence of clinical symptoms, physical or radiographic findings).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: a. subjects with type I diabetes, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible b. subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses 10 mg of prednisone or equivalent per day.
* Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association classification class > II), or serious cardiac arrhythmia.
* Clinically relevant diseases (for example, inflammatory bowel disease) and /or uncontrolled medical conditions, which, in the opinion of the investigator, might impair the subject's tolerance or ability to participate in the trial.
* Vaccine administration within 4 weeks of M7824 administration. Vaccination with live vaccines while on trial is prohibited. Administration of inactivated vaccines is allowed (for example, inactivated influenza vaccines).
* Pregnancy and breast feeding.
* History of conditions associated with bleeding diatheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of M7824 and radiation therapy in patients with metastatic HR+/HER2- breast cancer | 6 weeks after first administration of M7824
  Will be determined by dose limiting toxicity. RP2D defined as the highest dose level with no more than 1 patient with DLT out of 6 patients that are treated.
Safety and tolerability in patients with metastatic HR+/HER2- breast cancer | Start of study drug up to 30 days after study drug stopped
  Will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03. Recommended phase 2 dose (RP2D) will be determined by "3+3" design, and the recommended phase II dose is defined when 6 patients have been treated on that dose with no more than 1 dose limiting toxicity (DLT). DLT will be evaluated within 6 weeks after first administration of anti-PD-L1/TGFbetaRII fusion protein M7824 (M7824). Detailed information collected for each adverse event (AE) will include a description of the event, duration, severity, relationship to study treatment, action taken, and clinical outcome. Severity of AEs will be graded according to the CTCAE v 4.0. Summary of AEs will include only AEs that started or worsened during the on-treatment period, the treatment-emergent AEs. However, all safety data (including those from the pre- and post-treatment periods) will be listed and those collected during the pre- and post-treatment are to be flagged.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Start of study drug up to 90 days after study drug stopped
  PFS is defined as the time from treatment until objective tumor progression or death, whichever occurs first.
Overall survival (OS) | Start of study drug up to 90 days after study drug stopped
  OS is defined as the time from treatment until death from any cause.
Immunologic/molecular response | Up to 56 days
  Immunologic/molecular response is defined as % change in tumor infiltrating lymphocytes (TIL) pre and post therapy to M7824 and radiation therapy in patients with HR+/HER2- metastatic breast cancer.
Evaluation of the size of metastasis after treatment with M7824 with radiation (in-field) and non-irradiated (abscopal) sites | Up to 56 days
  Will be determined by Response Evaluation Criteria in Solid Tumors 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org